CLINICAL TRIAL: NCT05255978
Title: A Prospective/Retrospective, Observational Follow-up Study of Chronic Hepatitis B With Non-alcoholic Fatty Liver Disease.
Status: Recruiting | Type: Observational
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ20210524
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: the Effect of NAFLD on CHB

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective/retrospective, observational follow-up study of effects of fatty liver on chronic hepatitis B. Patients will join this study who undergo transient elastography with liver stiffness (LS) and CAP measurements or Ultrasonic examination. All recruited subjects will undergo comprehensive clinical, anthropometric and laboratory assessments at the time when transient elastography or Ultrasonic examination is performed. We plan to compare the relationship between chronic hepatitis B and non-alcoholic fatty liver disease. Patients will be divided into several groups based on the demand.

ELIGIBILITY:
Inclusion Criteria: age > 18 years, chronic hepatitis B patients -

Exclusion Criteria: patients with chronic hepatitis C or D and human immunodeficiency virus co-infection, excessive alcohol intake (≥30 g/d for men, ≥20 g/d for women), other chronic liver diseases (e.g. primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis, Wilson's disease), or on medications known to induce hepatic steatosis (including corticosteroids, methotrexate, and tamoxifen), and pregnancy.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age > 18 years chronic hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-02-24 (Estimated); Primary Completion 2023-06-24 (Estimated); Study Completion 2030-06-24 (Estimated)

PRIMARY OUTCOMES:
disease progression | 3 years to 10 years
  the effect of NAFLD on CHB

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China